CLINICAL TRIAL: NCT01479933
Title: Randomized Controlled Trial of Vitamin D Supplementation on Glucose Metabolism in Subjects With Components of the Metabolic Syndrome
Brief Title: Glucose Metabolism Effects of Vitamin D Supplementation in Prediabetes
Acronym: VitDmet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Academy of Finland (Other); Juho Vainio Foundation (Other); Finnish Foundation for Cardiovascular Research (Other); Diabetes Research Foundation, Finland (Other)
Responsible Party: Principal Investigator, Tomi-Pekka Tuomainen, Professor, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: VitDmet
Record Dates: First submitted 2011-08-29; First posted 2011-11-28 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Prediabetic State; Overweight; Obese
Keywords: vitamin D; cholecalciferol; supplementation; prediabetic state; obesity; glucose metabolism; gene expression; transcriptomics; epigenomics; immunological function; insulin sensitivity; peripheral mononuclear cells
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity; Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin D 40 (Experimental): Vitamin D3 40 micrograms (1600 IU) per day
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D 80 (Experimental): Vitamin D3 80 micrograms (3200 IU) per day
  Interventions: Dietary Supplement: Vitamin D 80
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 40 micrograms (1600 IU) per day
  Arms: Vitamin D 40
Dietary Supplement: Placebo — Inactive placebo
  Arms: Placebo
Dietary Supplement: Vitamin D 80 — Vitamin D3 80 micrograms (3200 IU) per day
  Arms: Vitamin D 80

SUMMARY:
Vitamin D deficiency is widespread throughout the world, and the deficiency has been associated with several chronic diseases, such as cardiovascular diseases and diabetes. In Nordic countries, like in Finland, there is a particular variation in vitamin D status, and during wintertime, when there is no exposure to ultraviolet-B light from the sun, serum concentrations of vitamin D decrease substantially. In Finland, some 40% of middle-aged men and one third of women also have some degree of impairment of glucose metabolism.

The purpose of this trial is to investigate the effects of two different daily doses of vitamin D on glucose metabolism in men 60 years of age or older and who are vitamin D deficient, have a high body mass index and at least two characteristics of cardio-metabolic syndrome.

Altogether 102 subjects with low serum calcidiol (<60 nmol/L) will be recruited and randomized to one of the three groups: 1) 40 µg/d vitamin D3, 2) 80 µg/d vitamin D3 or 3) placebo. The supplementation period will last for 6 months from September 2011 to March 2012.

The main hypotheses of the trial are: (1.) Vitamin D supplementation will improve glucose and insulin metabolism in people with a low baseline vitamin D status, in a dose-dependent manner. (2.) Vitamin D supplementation will have an effect on the expression of genes involved in glucose and insulin metabolism and inflammation. (3.) Vitamin D supplementation will have an effect on epigenetic changes in key genes participating in vitamin D metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Serum calcidiol <75 nmol/L
* Body mass index 25-35 kg/m2
* Impaired fasting glucose or impaired glucose tolerance (fasting glucose 5.6-7.0 mmol/L or 2h oral glucose tolerance test glucose 7.8-11.0 mmol/L)

Exclusion Criteria:

* Any chronic disease and condition, which may hamper to follow the intervention protocol (such as alcohol abuse)
* Any chronic disease or therapy which may mask or interact with the investigated effects (such as diabetes or systemic corticosteroid therapy)
* Any disease or state that raises a vitamin D related safety concern (such as chronic liver, thyroid or kidney disease, hypercalcemia, sarcoidosis or other granulomatous diseases such as active chronic tuberculosis or Wegener's granulomatosis)
* Use of supplements yielding vitamin D over 20 µg/d and unwillingness to discontinue the use.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Six months
  Change in insulin sensitivity measured by oral glucose tolerance test at baseline and after 6 months

SECONDARY OUTCOMES:
Peripheral blood mononuclear cell gene expression | Six months
Inflammation | Baseline to six months
  Change in inflammation measured as serum cytokines and adipose tissue inflammation at baseline and after 6 months
Adipose tissue gene expression | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Tomi-Pekka Tuomainen, MD, PhD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio Campus, Kuopio, Kuopio, Finland

REFERENCES:
- [Derived] Ryynanen J, Neme A, Tuomainen TP, Virtanen JK, Voutilainen S, Nurmi T, de Mello VD, Uusitupa M, Carlberg C. Changes in vitamin D target gene expression in adipose tissue monitor the vitamin D response of human individuals. Mol Nutr Food Res. 2014 Oct;58(10):2036-45. doi: 10.1002/mnfr.201400291. Epub 2014 Jul 28. PMID 24975273
- See also: University of Eastern Finland — http://www.uef.fi